CLINICAL TRIAL: NCT04548739
Title: Cerebral Autoregulation in Pediatric ECMO (ECMOX 2) : Autoregul ECMO - ECMOX2
Brief Title: Cerebral Autoregulation in Pediatric ECMO (ECMOX 2)
Acronym: ECMO-ECMOX2
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Istituto Giannina Gaslini (Other); Pediatric Intensive Care Unit, Trousseau University Hospital, France (Unknown); Pediatric Intensive Care Unit, Necker University Hospital, France (Unknown); Brain Physics Laboratory, Division of Neurosurgery, Department of Clinical Neurosciences, University of Cambridge, UK (Unknown)
Responsible Party: Sponsor
Other Study IDs: RC20_0066
Record Dates: First submitted 2020-06-04; First posted 2020-09-14 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS); Cardiogenic Shock; Cardiac Arrest
Keywords: ECMO; Cerebral autoregulation
MeSH Terms: conditions — Respiratory Distress Syndrome; Shock, Cardiogenic; Heart Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Children supported by Extra-Corporeal Membrane Oxygenation (ECMO) present a high risk of neurological complications and cerebral autoregulation (CA) impairment may be a risk factor. The first objective is to investigate the association between CA impairments and neurological outcome assessed by the onset of an ANE. The secondary objective is to study the underlying mechanisms influencing CA.

DETAILED DESCRIPTION:
Patients : All children treated by ECMO in the 4 PICUs involved in the study

Measurements : A correlation coefficient between the variations of regional cerebral oxygen saturation (rScO2) as a surrogate of cerebral blood flow and the variations of arterial blood pressure (ABP) is calculated as an index of autoregulation (cerebral oxygenation index (COx), ICM+ software®). CA is monitored either on left (COxl) or both sides. A COx > 0.3 is considered as critical. Neurological outcome is assessed by the onset of an acute neurologic event (ANE) during the ECMO run.

ELIGIBILITY:
Inclusion Criteria :

* Patients under the age of 18 years treated by ECMO

Exclusion Criteria :

* Lack of parental consent

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 100 children admitted to the Pediatric Intensive Care Unit (PICU) of Nantes (France), Trousseau (Paris, France), Necker (Paris, France) or Genoa (Italy) and supported by ECMO for hemodynamic or respiratory indication or during cardiac arrest resuscitation will be included in the study.
  As ECMO is an emergency procedure, emergency inclusions may be needed. Other observational study may be conducted in parallel in this population.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
Association between CA metrics and neurological outcome | 1 year
  Association between the percentage of time spent in critical region of CA and the onset of an acute neurological event (stroke and/or seizures and/or brain death) or not.

SECONDARY OUTCOMES:
Analysis of the influence of PCO2 on CA | 1 year
  Association between PCO2 value (mmHg) and COX value
Analysis of the influence of PCO2 on CA | 1 year
  Influence of ECMO settings on CA

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas JORAM, MD, Principal Investigator — Nantes University Hospital
Locations (4):
- France (3):
  - CHU de Nantes, Nantes
  - AP-HP Trousseau Hospital, Paris
  - AP-HP Necker Hospital, Paris
- Giannina Gaslini Institute (IRCCS), Genova, Italy

IPD SHARING:
Plan to Share IPD: Undecided